CLINICAL TRIAL: NCT05464966
Title: The Primary Objective of This Study Was to Investigate the Effect of Insulin on Myocardial Perfusion in Patients Undergoing Cardiac Surgery for CPB Using Transesophageal Echocardiography (TEE) to Detect CSBF and the Secondary Objective Was to Observe the Effect of Insulin on Cardiac Function and Markers of Myocardial Injury
Brief Title: The Primary Objective of This Study Was to Investigate the Effect of Insulin on Myocardial Perfusion and Cardiac Function in Patients Undergoing Cardiac Surgery for CPB Using Transesophageal Echocardiography (TEE) to Detect CSBF
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yangzhou University (Other)
Responsible Party: Principal Investigator, Zhuan Zhang, Principal Investigator, Yangzhou University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 20220515
Record Dates: First submitted 2022-05-15; First posted 2022-07-19 (Actual); Last update posted 2024-01-19 (Actual); Status verified 2024-01

CONDITIONS: Insulin
Keywords: Insulin; Perioperative period; Blood glucose; Heart protection
MeSH Terms: conditions — Insulin Resistance | interventions — glucose-insulin-potassium cardioplegic solution

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Glucose-insulin-potassium (Experimental)
  Interventions: Drug: Glucose insulin potassium
- Control (No Intervention)

INTERVENTIONS:
Drug: Glucose insulin potassium — After induction of anaesthesia,cardiac systolic-diastolic function was first measured by TEE, GIK solution was continuously pumped until the end of the procedure at a dose of 30 mU/kg/h of insulin, 0.12 g/kg/h of glucose and 0.06 mmol/kg/h of potassium chloride
  Arms: Glucose-insulin-potassium

SUMMARY:
The primary objective of this clinical trial was to investigate the effects of insulin on myocardial blood flow reflected by CSBF which was evaluated by TEE. The second aim was to observe the effect of insulin on cardiac function and markers of myocardial damage.

ELIGIBILITY:
Inclusion criteria included

1. age 55-80 years, ASA grade II-III, regardless of gender,
2. BMI 18.5-28.0 kg/m2,
3. scheduled for elective coronary artery bypass grafting (CABG), valve repair or replacement, or a combination of these procedures with cardiopulmonary bypass.

Exclusion criteria

1. non-first cardiac surgery;
2. emergency cardiac surgery;
3. severe heart failure with preoperative left ventricular ejection fraction <30%;
4. contraindication to TEE;
5. kidney disease requiring replacement therapy;
6. combined with multi-organ insufficiency;
7. Severe infection requiring continuous antibiotic treatment;
8. use of large doses of hormone or nonsteroidal anti-inflammatory drugs within the last 2 weeks.
9. after the patient entered the operating room, if the first blood glucose exceeded 180 mg/dl, a second test was performed 15 minutes later, and if the average of the two blood glucoses exceeded 180 mg/dl, the patient was excluded as well.

Elimination criteria included

1. unplanned secondary CPB;
2. need for intra-aortic balloon pump technical support during the study period;
3. TEE image acquired with poor quality.

Ages: 55 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 74 (Actual)
Dates: Start 2022-06-01 (Actual); Primary Completion 2023-05-31 (Actual); Study Completion 2023-06-30 (Actual)

PRIMARY OUTCOMES:
Changes in the coronary sinus blood flow spectrum | from 30 minutes after intubation to 1 hour after intubation , from 30minutes before the end of the surgery to the end of the surgery
  coronary sinus blood flow spectrum changes such as SVTI、DVTI、AVTI are assessed by TEE
Changes in left ventricular diastolic function | from 30 minutes after intubation to 1 hour after intubation , from 30minutes before the end of the surgery to the end of the surgery
  Changes in left ventricular diastolic function are assessed by TEE, such as changes in pulmonary venous blood flow

SECONDARY OUTCOMES:
Changes in the level of Systolic Blood Pressure/Diastolic Blood Pressure(Mean Arterial Pressure) | into ICU 30 minutes
  The above results should be measured immediately after induction, at the beginning of surgery, after administration of protamine, and at the end of surgery
Changes in the level of Cardiac output | into ICU 30 minutes
  The above results should be measured immediately after induction, at the beginning of surgery, after administration of protamine, and at the end of surgery
Changes in the level of Heart Rate | into ICU 30 minutes
  The above results should be measured immediately after induction, at the beginning of surgery, after administration of protamine, and at the end of surgery
Changes in the level of SVR | into ICU 30 minutes
  The above results should be measured immediately after induction, at the beginning of surgery, after administration of protamine, and at the end of surgery
Changes in the level of SVRI | into ICU 30 minutes
  The above results should be measured immediately after induction, at the beginning of surgery, after administration of protamine, and at the end of surgery
Changes in the level of Cardiac index | into ICU 30 minutes
  The above results should be measured immediately after induction, at the beginning of surgery, after administration of protamine, and at the end of surgery

CONTACTS AND LOCATIONS:
Locations (1):
- the Affiliated Hospital of Yangzhou University, Yangzhou University, Yangzhou, Jiangsu, China